CLINICAL TRIAL: NCT03934931
Title: Options for Delivering Isoniazid-Rifapentine (3HP) for TB Prevention: the 3HP Options Implementation Trial
Brief Title: Options for Delivering Isoniazid-Rifapentine (3HP) for TB Prevention (3HP Options Implementation Trial)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Makerere University (Other); Johns Hopkins Bloomberg School of Public Health (Other); University of Colorado, Denver (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01HL144406 (NIH); R01HL144406 (NIH)
Record Dates: First submitted 2019-04-22; First posted 2019-05-02 (Actual); Results first posted 2023-11-07 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Tuberculosis; Latent Tuberculosis; HIV/AIDS
Keywords: latent tuberculosis; tuberculosis; HIV/AIDS; implementation science; Uganda; 3HP; shared decision making; rifapentine
MeSH Terms: conditions — Tuberculosis; Latent Tuberculosis; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Facilitated Directly Observed Therapy (DOT) (Experimental): Facilitated DOT arm participants will attend the Mulago Immune Suppression Syndrome (ISS) clinic on a weekly basis to ingest 3HP medication under direct observation. DOT will be defined as a designated clinic staff member observing ingestion of each dose of 3HP. Additionally, participants randomized to facilitated DOT will receive: 1) DOT cards with instructions to present directly to the pharmacy for a pharmacy-only visit, without the need to wait in the general queue; 2) Automated short message service (SMS) or phone call reminders at no cost to participants the day before each appointment, 3) A fixed level of reimbursement (~$5/visit) for each weekly visit, conditional on either directly observed therapy or evidence of an adverse event that would preclude further treatment.
  Interventions: Other: Streamlined weekly DOT visits; Other: Weekly DOT visit reminders; Other: Cost reimbursement DOT
- Facilitated Self-Administered Therapy (SAT) (Experimental): Facilitated SAT participants will take their 1st dose of medication under direct observation and be given a 4-week 3HP supply to take weekly via self-administration. Participants will return to the Mulago ISS clinic after completing their 5th dose to review adherence data with the clinic pharmacy technician and receive 5 additional 3HP doses (doses 7-11). At the scheduled refill visit (dose 6) and end-of-treatment visit (dose 12) participants will ingest 3HP via direct observation. Participants will also receive: 1) Free automated SMS reminders or phone call reminders before each scheduled dose; 2) Weekly check-ins inquiring about side effects via two-way SMS with a follow-up phone call depending on participant response, 3) Fixed level of reimbursement (~$5/visit) for the refill/end-of-treatment visit, conditional on either directly observed therapy or evidence of an adverse event that would preclude further treatment.
  Interventions: Other: 99DOTS; Other: Weekly SAT dosing reminders/check-ins; Other: Cost reimbursement SAT
- Patient Choice between facilitated DOT and facilitated SAT (Experimental): Participants randomized to the Patient Choice between facilitated DOT and facilitated SAT arm will be offered a choice between arms 1 and 2. A research nurse will review each section of the decision aid with participants, discuss values and preferences, and, after addressing any questions, ask participants to select facilitated DOT or facilitated SAT. Participants will have the option to switch between DOT and SAT at any time. The reason for switching and time spent under each strategy will be recorded.
  Interventions: Other: Streamlined weekly DOT visits; Other: Weekly DOT visit reminders; Other: Cost reimbursement DOT; Other: 99DOTS; Other: Weekly SAT dosing reminders/check-ins; Other: Cost reimbursement SAT

INTERVENTIONS:
Other: Streamlined weekly DOT visits — Streamlined, weekly DOT clinic visits to have health worker observe medication ingestion and screen for side effects
  Arms: Facilitated Directly Observed Therapy (DOT); Patient Choice between facilitated DOT and facilitated SAT
Other: Weekly DOT visit reminders — Weekly SMS or interactive voice response (IVR) phone call reminder for DOT clinic visits
  Arms: Facilitated Directly Observed Therapy (DOT); Patient Choice between facilitated DOT and facilitated SAT
Other: Cost reimbursement DOT — Reimbursement of costs associated with weekly clinic visits (15,000 Ush/visit in Weeks 2-12)
  Arms: Facilitated Directly Observed Therapy (DOT); Patient Choice between facilitated DOT and facilitated SAT
Other: 99DOTS — 99DOTS-based digital adherence technology to monitor and promote adherence
  Arms: Facilitated Self-Administered Therapy (SAT); Patient Choice between facilitated DOT and facilitated SAT
Other: Weekly SAT dosing reminders/check-ins — Weekly SMS or IVR phone call dosing reminder/check-in for side effects
  Arms: Facilitated Self-Administered Therapy (SAT); Patient Choice between facilitated DOT and facilitated SAT
Other: Cost reimbursement SAT — Reimbursement of costs associated with streamlined refill and end-of treatment clinic visits (15,000 Ush/visit in Weeks 6 and 12)
  Arms: Facilitated Self-Administered Therapy (SAT); Patient Choice between facilitated DOT and facilitated SAT

SUMMARY:
The Options for Delivering Isoniazid-Rifapentine (3HP) for TB Prevention (3HP Options Implementation Trial) study will be a three-arm, open-label, parallel, randomized trial. This hybrid effectiveness-implementation trial will be conducted among people living with HIV infection (PLHIV) enrolled in HIV/AIDS care at the Mulago Immune Suppression Syndrome (i.e., HIV/AIDS) clinic in Kampala, Uganda. The overall objective of this study is to identify a patient-centered delivery strategy that will facilitate acceptance and completion of a three-month (12-dose) regimen of weekly rifapentine (RPT) and isoniazid (INH) by PLHIV enrolled in routine HIV/AIDS care in a high HIV/TB burden country. The primary outcome will be acceptance and completion of 3HP. Additional objectives will be to evaluate the implementation and cost-effectiveness of each delivery strategy.

DETAILED DESCRIPTION:
The overall objective of this study is to identify a patient-centered strategy that will facilitate 3HP uptake by PLHIV in the context of routine HIV/AIDS care in a high HIV/TB burden country. The investigators' central hypothesis is that offering PLHIV an informed choice between directly observed therapy (DOT) and self-administered therapy (SAT) delivery strategies that are optimized to overcome key barriers to treatment adherence will result in greater acceptance and completion of 3HP. To test this hypothesis, the investigators will conduct a pragmatic randomized trial of three optimized strategies for delivering 3HP. Eligible participants will be randomized to one of three arms to receive latent tuberculosis infection (LTBI) treatment with once weekly INH and RPT for 12 weeks given by either facilitated DOT, facilitated SAT, or an informed choice between facilitated DOT and facilitated SAT (with the assistance of a decision aid tool).

Primary Objective: To compare the uptake of 3HP under three delivery strategies: 1) Facilitated DOT; 2) Facilitated SAT; and 3) Informed patient choice (using a decision aid) between facilitated DOT and facilitated SAT. The primary outcome will be defined as the proportion of eligible participants who accept treatment and take at least 11 of 12 doses of RPT/INH within 16 weeks of treatment initiation. Study staff will assess medication dosing using clinic records for participants taking 3HP by DOT and using a combination of 99DOTS (Everwell Health Solutions, India) digital medication adherence technology records and pill counts at refill visits for participants taking 3HP by SAT.

Secondary Objectives:

1. To estimate the costs and compare the cost-effectiveness of the three strategies for delivering 3HP.
2. To identify processes and contextual factors that influence patient acceptance and completion of 3HP under each delivery strategy.
3. To identify clinic-level barriers to adoption and implementation of 3HP under each delivery strategy.
4. To determine the proportion of patients for whom 3HP treatment is discontinued due to adverse events/intolerance.
5. To determine the cumulative 16-month incidence of active TB in each arm, categorized as definite (positive sputum Xpert MTB/RIF or culture) or probable (TB medications started at the discretion of a clinician, with evidence of subsequent improvement).
6. To determine the cumulative 28-month incidence of active TB in each arm, categorized as definite (positive sputum Xpert MTB/RIF or culture) or probable (TB medications started at the discretion of a clinician, with evidence of subsequent improvement).

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive client engaged in care at the Mulago ISS clinic
* Weight ≥40kg
* Age 18 years or older
* Capacity to provide informed consent in English or Luganda

Exclusion Criteria:

* Suspicion of active TB based on positive World Health Organization (WHO) symptom screen AND elevated point-of-care (POC) C-reactive protein (CRP), or current or planned TB treatment
* Actively taking an antiretroviral medication contraindicated for use with rifapentine under contemporary WHO or Ugandan policy
* Contact of a TB patient with known resistance to isoniazid or rifamycins
* Women who are pregnant, breast feeding or intending to get pregnant in the next 120 days
* Prisoners
* Previously completed treatment for active TB or at least 6 months of isoniazid preventive therapy within past 2 years
* Not intending to remain within 25 km of the Mulago ISS clinic during the study period or to receive further care at the Mulago ISS clinic
* Lack of access to a mobile telephone or lack of willingness to receive SMS reminders
* Pre-existing documentation of clinical liver disease.
* History of sensitivity or intolerance to isoniazid or rifamycins
* Another household member already enrolled in the study (household members cannot be effectively randomized to different arms)
* Actively taking medication contraindicated for use with rifamycin (e.g., warfarin, phenytoin)

Mixed methods and health economic sub-studies will include a subset of participants enrolled in the trial, as well as clinic administrators and clinicians (clinical officer, doctor, nurse or pharmacist) involved in 3HP delivery at the Mulago ISS clinic.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1656 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2022-09-29 (Actual); Study Completion 2025-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adithya Cattamanchi, MD, Principal Investigator — University of California, San Francisco; David W Dowdy, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Mulago Immune Suppression Syndrome (ISS) Clinic, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Provided upon request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] TEMPRANO ANRS 12136 Study Group; Danel C, Moh R, Gabillard D, Badje A, Le Carrou J, Ouassa T, Ouattara E, Anzian A, Ntakpe JB, Minga A, Kouame GM, Bouhoussou F, Emieme A, Kouame A, Inwoley A, Toni TD, Ahiboh H, Kabran M, Rabe C, Sidibe B, Nzunetu G, Konan R, Gnokoro J, Gouesse P, Messou E, Dohoun L, Kamagate S, Yao A, Amon S, Kouame AB, Koua A, Kouame E, Ndri Y, Ba-Gomis O, Daligou M, Ackoundze S, Hawerlander D, Ani A, Dembele F, Kone F, Guehi C, Kanga C, Koule S, Seri J, Oyebi M, Mbakop N, Makaila O, Babatunde C, Babatounde N, Bleoue G, Tchoutedjem M, Kouadio AC, Sena G, Yededji SY, Assi R, Bakayoko A, Mahassadi A, Attia A, Oussou A, Mobio M, Bamba D, Koman M, Horo A, Deschamps N, Chenal H, Sassan-Morokro M, Konate S, Aka K, Aoussi E, Journot V, Nchot C, Karcher S, Chaix ML, Rouzioux C, Sow PS, Perronne C, Girard PM, Menan H, Bissagnene E, Kadio A, Ettiegne-Traore V, Moh-Semde C, Kouame A, Massumbuko JM, Chene G, Dosso M, Domoua SK, N'Dri-Yoman T, Salamon R, Eholie SP, Anglaret X. A Trial of Early Antiretrovirals and Isoniazid Preventive Therapy in Africa. N Engl J Med. 2015 Aug 27;373(9):808-22. doi: 10.1056/NEJMoa1507198. Epub 2015 Jul 20. PMID 26193126
- [Background] Dye C, Glaziou P, Floyd K, Raviglione M. Prospects for tuberculosis elimination. Annu Rev Public Health. 2013;34:271-86. doi: 10.1146/annurev-publhealth-031912-114431. Epub 2012 Dec 14. PMID 23244049
- [Background] Getahun H, Granich R, Sculier D, Gunneberg C, Blanc L, Nunn P, Raviglione M. Implementation of isoniazid preventive therapy for people living with HIV worldwide: barriers and solutions. AIDS. 2010 Nov;24 Suppl 5:S57-65. doi: 10.1097/01.aids.0000391023.03037.1f. No abstract available. PMID 21079430
- [Background] Namuwenge PM, Mukonzo JK, Kiwanuka N, Wanyenze R, Byaruhanga R, Bissell K, Zachariah R. Loss to follow up from isoniazid preventive therapy among adults attending HIV voluntary counseling and testing sites in Uganda. Trans R Soc Trop Med Hyg. 2012 Feb;106(2):84-9. doi: 10.1016/j.trstmh.2011.10.015. Epub 2011 Dec 10. PMID 22154974
- [Background] Martinson NA, Barnes GL, Moulton LH, Msandiwa R, Hausler H, Ram M, McIntyre JA, Gray GE, Chaisson RE. New regimens to prevent tuberculosis in adults with HIV infection. N Engl J Med. 2011 Jul 7;365(1):11-20. doi: 10.1056/NEJMoa1005136. PMID 21732833
- [Background] Sterling TR, Villarino ME, Borisov AS, Shang N, Gordin F, Bliven-Sizemore E, Hackman J, Hamilton CD, Menzies D, Kerrigan A, Weis SE, Weiner M, Wing D, Conde MB, Bozeman L, Horsburgh CR Jr, Chaisson RE; TB Trials Consortium PREVENT TB Study Team. Three months of rifapentine and isoniazid for latent tuberculosis infection. N Engl J Med. 2011 Dec 8;365(23):2155-66. doi: 10.1056/NEJMoa1104875. PMID 22150035
- [Background] Podany AT, Bao Y, Swindells S, Chaisson RE, Andersen JW, Mwelase T, Supparatpinyo K, Mohapi L, Gupta A, Benson CA, Kim P, Fletcher CV; AIDS Clinical Trials Group A5279 Study Team. Efavirenz Pharmacokinetics and Pharmacodynamics in HIV-Infected Persons Receiving Rifapentine and Isoniazid for Tuberculosis Prevention. Clin Infect Dis. 2015 Oct 15;61(8):1322-7. doi: 10.1093/cid/civ464. Epub 2015 Jun 16. PMID 26082504
- [Background] Weiner M, Egelund EF, Engle M, Kiser M, Prihoda TJ, Gelfond JA, Mac Kenzie W, Peloquin CA. Pharmacokinetic interaction of rifapentine and raltegravir in healthy volunteers. J Antimicrob Chemother. 2014 Apr;69(4):1079-85. doi: 10.1093/jac/dkt483. Epub 2013 Dec 15. PMID 24343893
- [Background] Swindells S, Ramchandani R, Gupta A, Benson CA, Leon-Cruz J, Mwelase N, Jean Juste MA, Lama JR, Valencia J, Omoz-Oarhe A, Supparatpinyo K, Masheto G, Mohapi L, da Silva Escada RO, Mawlana S, Banda P, Severe P, Hakim J, Kanyama C, Langat D, Moran L, Andersen J, Fletcher CV, Nuermberger E, Chaisson RE; BRIEF TB/A5279 Study Team. One Month of Rifapentine plus Isoniazid to Prevent HIV-Related Tuberculosis. N Engl J Med. 2019 Mar 14;380(11):1001-1011. doi: 10.1056/NEJMoa1806808. PMID 30865794
- [Background] Belknap R, Holland D, Feng PJ, Millet JP, Cayla JA, Martinson NA, Wright A, Chen MP, Moro RN, Scott NA, Arevalo B, Miro JM, Villarino ME, Weiner M, Borisov AS; TB Trials Consortium iAdhere Study Team. Self-administered Versus Directly Observed Once-Weekly Isoniazid and Rifapentine Treatment of Latent Tuberculosis Infection: A Randomized Trial. Ann Intern Med. 2017 Nov 21;167(10):689-697. doi: 10.7326/M17-1150. Epub 2017 Nov 7. PMID 29114781
- [Background] Liu X, Blaschke T, Thomas B, De Geest S, Jiang S, Gao Y, Li X, Buono EW, Buchanan S, Zhang Z, Huan S. Usability of a Medication Event Reminder Monitor System (MERM) by Providers and Patients to Improve Adherence in the Management of Tuberculosis. Int J Environ Res Public Health. 2017 Sep 25;14(10):1115. doi: 10.3390/ijerph14101115. PMID 28946683
- [Background] Institute of Medicine (US) Committee on Quality of Health Care in America. Crossing the Quality Chasm: A New Health System for the 21st Century. Washington (DC): National Academies Press (US); 2001. Available from http://www.ncbi.nlm.nih.gov/books/NBK222274/ PMID 25057539
- [Background] Charles C, Gafni A, Whelan T. Shared decision-making in the medical encounter: what does it mean? (or it takes at least two to tango). Soc Sci Med. 1997 Mar;44(5):681-92. doi: 10.1016/s0277-9536(96)00221-3. PMID 9032835
- [Background] Joosten EA, DeFuentes-Merillas L, de Weert GH, Sensky T, van der Staak CP, de Jong CA. Systematic review of the effects of shared decision-making on patient satisfaction, treatment adherence and health status. Psychother Psychosom. 2008;77(4):219-26. doi: 10.1159/000126073. Epub 2008 Apr 16. PMID 18418028
- [Background] Stacey D, Legare F, Lewis K, Barry MJ, Bennett CL, Eden KB, Holmes-Rovner M, Llewellyn-Thomas H, Lyddiatt A, Thomson R, Trevena L. Decision aids for people facing health treatment or screening decisions. Cochrane Database Syst Rev. 2017 Apr 12;4(4):CD001431. doi: 10.1002/14651858.CD001431.pub5. PMID 28402085
- [Background] Epstein RM, Franks P, Fiscella K, Shields CG, Meldrum SC, Kravitz RL, Duberstein PR. Measuring patient-centered communication in patient-physician consultations: theoretical and practical issues. Soc Sci Med. 2005 Oct;61(7):1516-28. doi: 10.1016/j.socscimed.2005.02.001. Epub 2005 Apr 15. PMID 16005784
- [Background] Durand MA, Carpenter L, Dolan H, Bravo P, Mann M, Bunn F, Elwyn G. Do interventions designed to support shared decision-making reduce health inequalities? A systematic review and meta-analysis. PLoS One. 2014 Apr 15;9(4):e94670. doi: 10.1371/journal.pone.0094670. eCollection 2014. PMID 24736389
- [Background] O'Connor AM, Rostom A, Fiset V, Tetroe J, Entwistle V, Llewellyn-Thomas H, Holmes-Rovner M, Barry M, Jones J. Decision aids for patients facing health treatment or screening decisions: systematic review. BMJ. 1999 Sep 18;319(7212):731-4. doi: 10.1136/bmj.319.7212.731. PMID 10487995
- [Background] Marseille E, Larson B, Kazi DS, Kahn JG, Rosen S. Thresholds for the cost-effectiveness of interventions: alternative approaches. Bull World Health Organ. 2015 Feb 1;93(2):118-24. doi: 10.2471/BLT.14.138206. Epub 2014 Dec 15. PMID 25883405
- [Background] Oxlade O, Schwartzman K, Benedetti A, Pai M, Heymann J, Menzies D. Developing a tuberculosis transmission model that accounts for changes in population health. Med Decis Making. 2011 Jan-Feb;31(1):53-68. doi: 10.1177/0272989X10369001. Epub 2010 Jun 2. PMID 20519452
- [Background] Dowdy DW, Rodriguez RM, Hare CB, Kaplan B. Cost-effectiveness of targeted human immunodeficiency virus screening in an urban emergency department. Acad Emerg Med. 2011 Jul;18(7):745-53. doi: 10.1111/j.1553-2712.2011.01110.x. PMID 21762236
- [Background] Samandari T, Agizew TB, Nyirenda S, Tedla Z, Sibanda T, Shang N, Mosimaneotsile B, Motsamai OI, Bozeman L, Davis MK, Talbot EA, Moeti TL, Moffat HJ, Kilmarx PH, Castro KG, Wells CD. 6-month versus 36-month isoniazid preventive treatment for tuberculosis in adults with HIV infection in Botswana: a randomised, double-blind, placebo-controlled trial. Lancet. 2011 May 7;377(9777):1588-98. doi: 10.1016/S0140-6736(11)60204-3. Epub 2011 Apr 12. PMID 21492926
- [Background] Dowdy DW, Houben R, Cohen T, Pai M, Cobelens F, Vassall A, Menzies NA, Gomez GB, Langley I, Squire SB, White R; TB MAC meeting participants. Impact and cost-effectiveness of current and future tuberculosis diagnostics: the contribution of modelling. Int J Tuberc Lung Dis. 2014 Sep;18(9):1012-8. doi: 10.5588/ijtld.13.0851. PMID 25189546
- [Background] Menzies NA, Cohen T, Lin HH, Murray M, Salomon JA. Population health impact and cost-effectiveness of tuberculosis diagnosis with Xpert MTB/RIF: a dynamic simulation and economic evaluation. PLoS Med. 2012;9(11):e1001347. doi: 10.1371/journal.pmed.1001347. Epub 2012 Nov 20. PMID 23185139
- [Background] Sandelowski M, Leeman J. Writing usable qualitative health research findings. Qual Health Res. 2012 Oct;22(10):1404-13. doi: 10.1177/1049732312450368. Epub 2012 Jun 28. PMID 22745362
- [Background] Sandelowski MJ. Justifying qualitative research. Res Nurs Health. 2008 Jun;31(3):193-5. doi: 10.1002/nur.20272. No abstract available. PMID 18288640
- [Background] Voils CI, Sandelowski M, Barroso J, Hasselblad V. Making Sense of Qualitative and Quantitative Findings in Mixed Research Synthesis Studies. Field methods. 2008;20(1):3-25. doi: 10.1177/1525822X07307463. PMID 18677415
- [Background] Spiegelman D, Hertzmark E. Easy SAS calculations for risk or prevalence ratios and differences. Am J Epidemiol. 2005 Aug 1;162(3):199-200. doi: 10.1093/aje/kwi188. Epub 2005 Jun 29. No abstract available. PMID 15987728
- [Derived] Kadota JL, Musinguzi A, Aschmann HE, Akello L, Welishe F, Nakimuli J, Berger CA, Kiwanuka N, Phillips PPJ, Katamba A, Dowdy DW, Cattamanchi A, Semitala FC. Adverse Events Reported During Weekly Isoniazid-Rifapentine (3HP) Tuberculosis Preventive Treatment Among People With Human Immunodeficiency Virus in Uganda. Open Forum Infect Dis. 2024 Nov 14;11(11):ofae667. doi: 10.1093/ofid/ofae667. eCollection 2024 Nov. PMID 39582503
- [Derived] Musinguzi A, Kasidi JR, Kadota JL, Welishe F, Nakitende A, Akello L, Nakimuli J, Kunihira LT, Opira B, Baik Y, Patel D, Sammann A, Berger CA, Aschmann HE, Nahid P, Belknap R, Kamya MR, Handley MA, Phillips PPJ, Kiwanuka N, Katamba A, Dowdy DW, Cattamanchi A, Semitala FC, Katahoire AR. Evaluating the implementation of weekly rifapentine-isoniazid (3HP) for tuberculosis prevention among people living with HIV in Uganda: A qualitative evaluation of the 3HP Options Trial. PLOS Glob Public Health. 2024 Oct 24;4(10):e0003347. doi: 10.1371/journal.pgph.0003347. eCollection 2024. PMID 39446746
- [Derived] Semitala FC, Kadota JL, Musinguzi A, Welishe F, Nakitende A, Akello L, Kunihira Tinka L, Nakimuli J, Ritar Kasidi J, Bishop O, Nakasendwa S, Baik Y, Patel D, Sammann A, Nahid P, Belknap R, Kamya MR, Handley MA, Phillips PP, Katahoire A, Berger CA, Kiwanuka N, Katamba A, Dowdy DW, Cattamanchi A. Comparison of 3 optimized delivery strategies for completion of isoniazid-rifapentine (3HP) for tuberculosis prevention among people living with HIV in Uganda: A single-center randomized trial. PLoS Med. 2024 Feb 20;21(2):e1004356. doi: 10.1371/journal.pmed.1004356. eCollection 2024 Feb. PMID 38377166
- [Derived] Semitala FC, Kadota JL, Musinguzi A, Nabunje J, Welishe F, Nakitende A, Akello L, Bishop O, Patel D, Sammann A, Nahid P, Belknap R, Kamya MR, Handley MA, Phillips PPJ, Katahoire A, Berger CA, Kiwanuka N, Katamba A, Dowdy DW, Cattamanchi A. Completion of isoniazid-rifapentine (3HP) for tuberculosis prevention among people living with HIV: Interim analysis of a hybrid type 3 effectiveness-implementation randomized trial. PLoS Med. 2021 Dec 16;18(12):e1003875. doi: 10.1371/journal.pmed.1003875. eCollection 2021 Dec. PMID 34914696
- [Derived] Kadota JL, Musinguzi A, Nabunje J, Welishe F, Ssemata JL, Bishop O, Berger CA, Patel D, Sammann A, Katahoire A, Nahid P, Belknap R, Phillips PPJ, Namusobya J, Kamya M, Handley MA, Kiwanuka N, Katamba A, Dowdy D, Semitala FC, Cattamanchi A. Protocol for the 3HP Options Trial: a hybrid type 3 implementation-effectiveness randomized trial of delivery strategies for short-course tuberculosis preventive therapy among people living with HIV in Uganda. Implement Sci. 2020 Aug 12;15(1):65. doi: 10.1186/s13012-020-01025-8. PMID 32787925

RESULTS

PARTICIPANT FLOW:
Groups:
- Facilitated Directly Observed Therapy (DOT): Facilitated directly observed therapy (DOT) arm participants will attend the Mulago Immune Suppression Syndrome (ISS) clinic on a weekly basis to ingest 3HP medication under direct observation. DOT will be defined as a designated clinic staff member observing ingestion of each dose of 3HP. Additionally, participants randomized to facilitated DOT will receive: 1) DOT cards with instructions to present directly to the pharmacy for a pharmacy-only visit, without the need to wait in the general queue; 2) Automated short message service (SMS) or phone call reminders at no cost to participants the day before each appointment, 3) A fixed level of reimbursement (~$5/visit) for each weekly visit, conditional on either directly observed therapy or evidence of an adverse event that would preclude further treatment.
  Streamlined weekly DOT visits: Streamlined, weekly DOT clinic visits to have health worker observe medication ingestion and screen for side effects
  Weekly DOT visit reminders: Weekly SMS or interactive voice response (IVR) phone call reminder for DOT clinic visits
  Cost reimbursement DOT: Reimbursement of costs associated with weekly clinic visits (15,000 Ush/visit in Weeks 2-12)
- Facilitated Self-Administered Therapy (SAT): Facilitated self-administered therapy (SAT) participants will take their 1st dose of medication under direct observation and be given a 4-week 3HP supply to take weekly via self-administration. Participants will return to the Mulago ISS clinic after completing their 5th dose to review adherence data with the clinic pharmacy technician and receive 5 additional 3HP doses (doses 7-11). At the scheduled refill visit (dose 6) and end-of-treatment visit (dose 12) participants will ingest 3HP via direct observation. Participants will also receive: 1) Free automated SMS reminders or phone call reminders before each scheduled dose; 2) Weekly check-ins inquiring about side effects via two-way SMS with a follow-up phone call depending on participant response, 3) Fixed level of reimbursement (~$5/visit) for the refill/end-of-treatment visit, conditional on either directly observed therapy or evidence of an adverse event that would preclude further treatment.
  99DOTS: 99DOTS-based digital adherence technology to monitor and promote adherence
  Weekly SAT dosing reminders/check-ins: Weekly SMS or IVR phone call dosing reminder/check-in for side effects
  Cost reimbursement SAT: Reimbursement of costs associated with streamlined refill and end-of treatment clinic visits (15,000 Ush/visit in Weeks 6 and 12)
Period: Overall Study
Arm/Group | Facilitated Directly Observed Therapy (DOT) | Facilitated Self-Administered Therapy (SAT) | Patient Choice Between Facilitated DOT and Facilitated SAT
Started | 552 | 552 | 552 (Participant Choice between Facilitated DOT and Facilitated SAT was not split up to separately describe the number of participants who received each treatment regiment because the Participant Choice arm was analyzed as a single arm in the primary analysis.)
Completed | 551 | 552 | 552
Not Completed | 1 | 0 | 0
Not completed — Excluded as a duplicate enrollment | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 1 participant in the DOT arm was excluded as a duplicate enrollment
Groups:
- Total: Total of all reporting groups
Arm/Group | Facilitated Directly Observed Therapy (DOT) | Facilitated Self-Administered Therapy (SAT) | Patient Choice Between Facilitated DOT and Facilitated SAT | Total
Number analyzed (Participants) | 551 | 552 | 552 | 1655
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 42 [36 to 48] | 42 [36 to 48] | 42 [36 to 48] | 42 [36 to 48]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 378 | 375 | 369 | 1122
  Male | 173 | 177 | 183 | 533
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 551 | 552 | 552 | 1655
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Uganda | 551 | 552 | 552 | 1655
Prior Tuberculosis [Count of Participants; unit: Participants] | 104 | 108 | 89 | 301
Time on Antiretroviral therapy (ART) [Median (Inter-Quartile Range); unit: years] | 9.0 [5.8 to 12.4] | 9.1 [5.6 to 12.5] | 9.1 [5.5 to 12.7] | 9.0 [5.6 to 12.5]

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Who Accepted and Completed 3HP
Description: The count of eligible participants who accept treatment and take at least 11 of 12 once weekly doses of rifapentine (RPT)/isoniazid (INH) within 16 weeks of treatment initiation divided by the count of those randomized.
Time Frame: Within 16 weeks of treatment initiation
Population: 1,656 people were eligible and randomized. One participant was erroneously re-randomized (facilitated DOT arm) after an initial enrollment; data from their second randomization was excluded. 1,655 were included in the primary outcome analysis.
Measure: Number; unit: proportion of participants
Arm/Group | Facilitated Directly Observed Therapy (DOT) | Facilitated Self-Administered Therapy (SAT) | Patient Choice Between Facilitated DOT and Facilitated SAT
Number analyzed (Participants) | 551 | 552 | 552
proportion of participants | 0.946 | 0.922 | 0.944

2. Secondary Outcome: Proportion of Participants Who Accepted 3HP Treatment
Description: The count of eligible people living with HIV (PLHIV) offered 3HP who accept to initiate treatment (by age, gender, CD4 stratum, viral load suppression) divided by the count of those randomized.
Time Frame: Within 16 weeks of treatment initiation
Population: 1,656 people were eligible and randomized. One participant was erroneously re-randomized (facilitated DOT arm) after an initial enrollment; data from their second randomization was excluded. 1,655 were included in this secondary outcome analysis.
Measure: Number; unit: proportion of participants
Arm/Group | Facilitated Directly Observed Therapy (DOT) | Facilitated Self-Administered Therapy (SAT) | Patient Choice Between Facilitated DOT and Facilitated SAT
Number analyzed (Participants) | 551 | 552 | 552
proportion of participants | 0.998 | 1.00 | 0.995

3. Secondary Outcome: Proportion of Participants Who Completed 3HP Treatment
Description: Count of participants who take at least 11 of 12 doses within 16 weeks of treatment initiation divided by the count those who take at least one dose of 3HP.
Time Frame: Within 16 weeks of treatment initiation
Population: Those analyzed included the number of participants who took at least one dose of 3HP.
Measure: Number; unit: proportion of participants
Arm/Group | Facilitated Directly Observed Therapy (DOT) | Facilitated Self-Administered Therapy (SAT) | Patient Choice Between Facilitated DOT and Facilitated SAT
Number analyzed (Participants) | 550 | 552 | 549
proportion of participants | 0.947 | 0.922 | 0.949

4. Secondary Outcome: Proportion of People Who Discontinued 3HP Treatment Due to Adverse Events/Intolerance
Description: Count of participants for whom treatment is discontinued due to adverse events or intolerance divided by the count of those who initiated 3HP.
Time Frame: Within 16 weeks of treatment initiation
Population: Those analyzed included the number of participants who took at least one dose of 3HP.
Measure: Number; unit: proportion of participants
Arm/Group | Facilitated Directly Observed Therapy (DOT) | Facilitated Self-Administered Therapy (SAT) | Patient Choice Between Facilitated DOT and Facilitated SAT
Number analyzed (Participants) | 550 | 552 | 549
proportion of participants | 0.0054 | 0.013 | 0.0073

5. Secondary Outcome: Cumulative Incidence of Tuberculosis (TB)
Description: Cumulative 16-month incidence of active TB in each arm
Time Frame: from date of 3HP treatment completion (11/12 doses) or once reached 16 weeks (regardless of number of doses taken) until time of active TB diagnosis or treatment initiation, death, loss to follow-up or end of the 12-month post-treatment follow-up period
Reporting Status: Not Posted

6. Secondary Outcome: Cumulative Incidence of TB
Description: Cumulative 28-month incidence of active TB in each arm
Time Frame: from date of 3HP treatment completion (11/12 doses) or once reached 16 weeks (regardless of number of doses taken) until time of active TB diagnosis or treatment initiation, death, loss to follow-up or end of the 24-month post-treatment follow-up period
Reporting Status: Not Posted

7. Secondary Outcome: Cost Effectiveness (Patient Perspective)
Description: The incremental patient cost per disability-adjusted life year (DALY) averted.
Time Frame: At the conclusion of the study period, estimated 3 years
Reporting Status: Not Posted

8. Secondary Outcome: Cost Effectiveness (Health System Perspective)
Description: The incremental health system cost per disability-adjusted life year (DALY) averted.
Time Frame: At the conclusion of the study period, estimated 3 years
Reporting Status: Not Posted

9. Secondary Outcome: Cost Effectiveness (Overall Perspective)
Description: Incremental cost of each delivery strategy per disability adjusted life year (DALY) averted.
Time Frame: At the conclusion of the study period, estimated 3 years
Reporting Status: Not Posted

10. Secondary Outcome: Visit Cost Reimbursement - Overall
Description: Proportion reimbursed overall
Time Frame: Through study completion, an average of 16 weeks
Reporting Status: Not Posted

11. Secondary Outcome: Visit Cost Reimbursement
Description: Proportion reimbursed on the same day as each 3HP clinic visit
Time Frame: On the same day as each 3HP clinic visit throughout study completion, an average of 16 weeks
Reporting Status: Not Posted

12. Secondary Outcome: Time to Complete Clinic Visit - Mean Minutes
Description: Mean number of minutes for each DOT/refill visit
Time Frame: On the same day as each 3HP clinic visit throughout study completion, an average of 16 weeks
Reporting Status: Not Posted

13. Secondary Outcome: Time to Complete Clinic Visit - Median Minutes
Description: Median number of minutes for each DOT/refill visit
Time Frame: On the same day as each 3HP clinic visit throughout study completion, an average of 16 weeks
Reporting Status: Not Posted

14. Secondary Outcome: Short Messages Service (SMS) or Interactive Voice Response (IVR) Phone Call Reminders Delivered - Clinic Visits
Description: Proportion of SMS or IVR phone call reminders delivered to participants for clinic visits
Time Frame: The day before each 3HP clinic visit throughout study completion, an average of 16 weeks
Reporting Status: Not Posted

15. Secondary Outcome: Screening for Active TB
Description: Proportion of participants screened for active TB during DOT or refill visits
Time Frame: On the same day as each 3HP clinic visit throughout study completion, an average of 16 weeks
Reporting Status: Not Posted

16. Secondary Outcome: Screening for Side Effects
Description: Proportion of participants screened for side effects during DOT or refill visits.
Time Frame: On the same day as each 3HP clinic visit throughout study completion, an average of 16 weeks
Reporting Status: Not Posted

17. Secondary Outcome: Dosing Confirmation Via 99DOTS (SAT Only)
Description: Proportion of doses confirmed using digital adherence technology. Doses directly observed (i.e., during initial or refill visits) will not be included in the denominator.
Time Frame: On the same day as each scheduled dose throughout study completion, an average of 16 weeks
Reporting Status: Not Posted

18. Secondary Outcome: SMS or IVR Phone Call Reminders Delivered - Medication Dosing (SAT Only)
Description: Proportion of SMS or IVR phone call reminders delivered to participants for medication dosing
Time Frame: The day before each scheduled dose throughout study completion, an average of 16 weeks
Reporting Status: Not Posted

19. Secondary Outcome: SMS or IVR Phone Calls Delivered - Weekly check-in (SAT Only)
Description: Proportion of weekly SMS or IVR phone call check-ins delivered to participants
Time Frame: On the same day as each scheduled dose throughout study completion, an average of 16 weeks
Reporting Status: Not Posted

20. Secondary Outcome: SMS or IVR Phone Call Reminders Delivered - Missed Dose (SAT Only)
Description: Proportion of SMS or IVR phone call reminders delivered to participants following missed doses
Time Frame: 24 hours after missed scheduled dose throughout study completion, an average of 16 weeks
Reporting Status: Not Posted

21. Secondary Outcome: SMS or IVR Phone Call Missed Appointment Reminders Delivered
Description: Proportion of SMS or IVR phone call reminders delivered to participants following missed appointments
Time Frame: 24 hours after missed scheduled appointment throughout study completion, an average of 16 weeks
Reporting Status: Not Posted

22. Secondary Outcome: Follow up (Phone Calls or Home Visits) for Negative Response to Weekly SMS or IVR Phone Call check-in (SAT Only)
Description: Proportion of participants who receive appropriate follow-up (phone call or home visit) for lack of response/negative response to weekly check-in SMS or IVR phone call
Time Frame: 24 hours after negative response throughout study completion, an average of 16 weeks
Reporting Status: Not Posted

23. Secondary Outcome: Costs of Preventive Services
Description: Mean total participant costs related to TB preventive care services
Time Frame: Through study completion, an average of 16 weeks
Reporting Status: Not Posted

24. Secondary Outcome: Participant Satisfaction
Description: Mean score on participant satisfaction questionnaire
Time Frame: Through study completion, an average of 16 weeks
Reporting Status: Not Posted

25. Secondary Outcome: Barriers to 3HP Delivery From the Provider/Clinic Perspective
Description: Thematic interpretation of provider- and clinic-level barriers to care from provider focus group discussions.
Time Frame: At the conclusion of the study period, estimated 3 years
Reporting Status: Not Posted

26. Secondary Outcome: Barriers to 3HP Completion From the Patient Perspective
Description: Thematic interpretation of barriers to 3HP completion from patient interviews
Time Frame: Through study completion, an average of 16 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected weekly over the course of 3HP treatment duration (up to 16 weeks after treatment initiation)
Description: Adverse Events (AE) pre-specified to be reported according to participant randomization; AEs were not reported with respect to the specific intervention received by the participant in the "Patient Choice Between Facilitated DOT and Facilitated SAT" Arm, only the randomization group.
  Facilitated DOT: weekly in-person by pharmacy technician using standard checklist. Facilitated SAT: dose 2-5 & 7-11: two-way interactive voice response phone calls; dose 6 & 12: in-person using standard checklist
Arm/Group | Facilitated Directly Observed Therapy (DOT) | Facilitated Self-Administered Therapy (SAT) | Patient Choice Between Facilitated DOT and Facilitated SAT
All-Cause Mortality (participants affected / at risk) | 1/551 | 0/552 | 0/552
Serious Adverse Events (participants affected / at risk) | 3/551 | 7/552 | 4/552
Other Adverse Events (participants affected / at risk) | 83/551 | 86/552 | 76/552
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Facilitated Directly Observed Therapy (DOT) (N=551) | Facilitated Self-Administered Therapy (SAT) (N=552) | Patient Choice Between Facilitated DOT and Facilitated SAT (N=552)
Generalized pruritus/skin rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Hearing impairment (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
3HP-related hypersensitivity (General disorders) | 0 (0) | 2 (2) | 0 (0)
Flu-like syndrome (General disorders) | 0 (0) | 1 (1) | 1 (1)
Toxic Conjunctivitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Venous thromboembolism (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Facilitated Directly Observed Therapy (DOT) (N=551) | Facilitated Self-Administered Therapy (SAT) (N=552) | Patient Choice Between Facilitated DOT and Facilitated SAT (N=552)
Fever (General disorders) | 19 (21) | 21 (25) | 17 (19)
Headache (Nervous system disorders) | 23 (23) | 24 (29) | 16 (16)
Weakness (General disorders) | 20 (20) | 20 (21) | 14 (14)
Joint pain (Musculoskeletal and connective tissue disorders) | 21 (24) | 21 (26) | 29 (33)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-03-20): https://cdn.clinicaltrials.gov/large-docs/31/NCT03934931/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-26): https://cdn.clinicaltrials.gov/large-docs/31/NCT03934931/SAP_001.pdf
  • Informed Consent Form (2021-09-07): https://cdn.clinicaltrials.gov/large-docs/31/NCT03934931/ICF_002.pdf